CLINICAL TRIAL: NCT06265844
Title: A Randomly Controlled Study to Explore the Effect of Oral Feeding in Dysphagia for Nasopharyngeal Carcinoma
Brief Title: Multifunctional Nutrition Tube in Dysphagia for Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IOE-Biyanai
Record Dates: First submitted 2024-01-28; First posted 2024-02-20 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The observation group (Experimental): During the 15-day treatment, both groups of patients are hospitalized, while conventional care and enteral nutrition support are provided to the two groups. Specifically, conventional care includes health education, dietary adjustments, nasopharyngeal hygiene, management of risk factors (blood pressure and lipid control, etc.), exercise rehabilitation, and psychological support. The frequency and content of these interventions are arranged based on the patients; health condition. The observation group receives Intermittent Oro-esophageal Tube Feeding for enteral nutrition support
  Interventions: Device: Intermittent Oral-esophageal Tube Feeding; Behavioral: comprehensive rehabilitation therapy
- The control group (Active Comparator): During the 15-day treatment, both groups of patients are hospitalized, while conventional care and enteral nutrition support are provided to the two groups. Specifically, conventional care includes health education, dietary adjustments, nasopharyngeal hygiene, management of risk factors (blood pressure and lipid control, etc.), exercise rehabilitation, and psychological support. The frequency and content of these interventions are arranged based on the patients; health condition.The control group receives nasogastric tube for enteral nutrition support
  Interventions: Device: Nasogastric Tube Feeding; Behavioral: comprehensive rehabilitation therapy

INTERVENTIONS:
Device: Intermittent Oral-esophageal Tube Feeding — The specific procedure was as follows: the infant was placed in a semi-recumbent or sitting position with the head fixed. Before each feeding, the infant's oral and nasal secretions were to be cleared. An intermittent oro-esophageal tube was appropriately lubricated with water on the head part. The professional medical staff held the tube and slowly inserted it through one side of the mouth into the upper part of the esophagus. The depth of insertion depended on the patient's age and height. After each feeding, the tube was immediately removed, and the patient was held upright for at least 30 minutes in case of reflux.
  Arms: The observation group
Device: Nasogastric Tube Feeding — Nasogastric Tube Feeding were used for feeding to provide nutritional support. Each feeding was administered by a nurse using the infant's mother's breast milk through the tube. The amount of each feeding varied from 20 to 100 ml depending on the age of the infant, with feedings given every 2 to 3 hours, approximately 10 times per day. The duration of each feeding procedure ranged from 10 to 20 minutes. The total daily intake ranged from 200 to 1000 ml. Each tube was kept indwelling for 5 to 7 days. When the tube needed to be replaced, it was removed after the last feeding of a day and a new tube was to be inserted through the other nostril on the following morning to continue the nutritional support.
  Arms: The control group
Behavioral: comprehensive rehabilitation therapy — Both groups were given comprehensive rehabilitation therapy. The main intervention measures included: 1) non-invasive ventilator treatment, generally at least once every night and typically not exceeding continuous daily usage.; 2) attention to feeding and sleeping positions, with a recommended sleeping position of lateral recumbent and the head of the bed raised by 20-30°; 3) swallowing function training, such as tongue muscle stretching training, assisted anterior jaw protrusion training, lemon ice stimulation to the soft palate, pharyngeal wall, etc., generally 5 days per week, twice per day, 5-20 minutes each time; 4) pulmonary ultrashort wave therapy, generally at least 2-3 times a week, and not more than once a day; 5) physical therapy, such as intensive training for gross motor functions including lifting the head, turning over, sitting, crawling, standing, etc., generally 3-5 days per week, 1-2 times per day, 5-20 min each time.

SUMMARY:
This is a prospective multicenter study with patients with delayed dysphagia after radiotherapy for NPC. Patients enrolled are randomly divided equally into the observation group and the control group. All patients receive conventional care, and the observation group received IOE while the control group received NGT for enteral nutrition support. Baseline information (demographics, medical history, etc.), nutritional status at admission and after treatment, depression, dysphagia, and quality of life (QOL) after treatment as well as adverse events are compared.

DETAILED DESCRIPTION:
Palliation to delayed dysphagia after radiotherapy for nasopharyngeal carcinoma (NPC) continues to be a challenge. Although nasogastric tube feeding (NGT) has been adopted widely, the weaknesses have yet to be improved by another enteral nutrition support mode. This study aims to observe the clinical efficacy of intermittent oro-esophageal tube feeding (IOE) in the treatment of delayed dysphagia after radiotherapy for (NPC). This is a prospective multicenter study with patients with delayed dysphagia after radiotherapy for NPC. Patients enrolled are randomly divided equally into the observation group and the control group. All patients receive conventional care, and the observation group received IOE while the control group received NGT for enteral nutrition support. Baseline information (demographics, medical history, etc.), nutritional status at admission and after treatment, depression, dysphagia, and quality of life (QOL) after treatment as well as adverse events are compared.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* With the history of NPC and radiation therapy.
* With dysphagia occurred at least three years after radiotherapy (confirmed by videofluoroscopic swallowing study), in need of and feasible for enteral nutrition support.
* Conscious and with stable vital signs;
* Willing to participate and sign the written informed consent form either personally or by a family member.

Exclusion Criteria:

* Presence of other diseases that might cause dysphagia.
* With distant metastasis of tumors, or complicated with severe systemic disorders or malignancies.
* Concurrent participation in other treatments that could interfere with the trial.
* Inability to cooperate with treatment due to aphasia, mental health issues, etc.
* Received tube feeding for enteral nutrition support within the past three years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | day 1 and day 15
  Hemoglobin was recorded through the blood routine test. (Hb, g/L)
Serum albumin | day 1 and day 15
  Serum albumin was recorded through the blood routine test. (ALB, g/L)
Body Mass Index | day 1 and day 15
  Body Mass Index was assessed with the combination of body weight and height: weight (kg)/ [height (m)] ^2
Serum prealbumin | day 1 and day 15
  Serum prealbumin was recorded through the blood routine test.(PA, g/L)

SECONDARY OUTCOMES:
Depression | day 1 and day 15
  The PATIENT HEALTH QUESTIONNAIRE scale is utilized to evaluate the depression of patients at admission and after treatment. Options representing varying degrees of severity, ranging from 0 to 3 were provided in each aspect. The total scores between 0 and 4 were classified as negative, indicating the absence of depressive symptoms, while scores above 4 were classified as positive, indicating the presence of potential depressive symptoms.
Functional Oral Intake Scale | day 1 and day 15
  The Functional Oral Intake Scale (FOIS) was used to evaluate function of oral intake. In the FOIS assessment, two professional rehabilitation therapists communicated with the patients, observed and recorded to assess their swallowing function. The assessment scale consists of seven levels, with a higher level indicating progressively better swallowing function (less dysphagia).
Penetration-Aspiration Scale | day 1 and day 15
  In this study, the Penetration-Aspiration Scale (PAS) was recruited, which was a commonly used to evaluate the occurrence of penetration or aspiration during swallowing. It categorizes dysphagia into eight levels, with Level 0 indicating no penetration or aspiration and Level 8 indicating severe aspiration. A higher level indicates more severe dysphagia.
Swallowing-Quality of Life questionnaire | day 1 and day 15
  The Chinese version of the Swallowing-Quality of Life questionnaire (SWAL-QOL) was used to assess the quality of life of patients.he Likert scale ranging from 1 to 5 was utilized for scoring, with a total of 44 items, including difficulties in swallowing, dietary restrictions, oral health, social communication, and others. The total score was converted to a standard percentage scale ranging from 0 to 100, with positively correlated with quality of life.
Feeding amount | day 1 and day 15
  The total amount of nutrients consumed by the patient on the day was recorded, excluding fresh water, units: milliliters

CONTACTS AND LOCATIONS:
Overall Officials: Qingfeng Tian, Doctor, Study Director — Zhengzhou University
Locations (1):
- Saint Martin Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No